CLINICAL TRIAL: NCT00529802
Title: An Exploratory Study Evaluating FDG-PET as a Predictive Marker for mTOR Directed Therapy With RAD001 in Metastatic Renal Cell Cancer
Brief Title: Exploratory Study Evaluating Fluorodeoxyglucose - Position Emission Tomography as a Predictive Marker for Therapy With RAD001 in Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15599B
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: metastatic; renal; cell; carcinoma; cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis; Carcinoma; Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus (RAD001) 10mg daily (Experimental): All patients were to receive 10mg everolimus (RAD001) daily.
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — take 2 tablets of RAD001 once a day by mouth (10 mg per day)

SUMMARY:
The purpose of this study is to learn if PET scanning can predict the degree of tumor shrinkage with the study drug RAD001 in subjects who have advanced renal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic renal cancer refractory to sorafenib or sunitinib therapy
* At least one measurable site of disease according to RECIST criteria that has not been previously irradiated.
* 18 years of age or older
* Minimum of two weeks since any major surgery, completion of radiation, or completion of all prior standard systemic anticancer therapy and adequately recovered from the acute toxicities of any prior therapy.
* World Health Organization (WHO) performance status <= 2
* Adequate bone marrow function
* Adequate liver function
* Adequate creatinine clearance
* Signed informed consent

Exclusion Criteria:

* Prior treatment with any investigational drug within the previous 4 weeks
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Patients who have a history of another primary malignancy ≤ 3 years, with the exceptions of non-melanoma skin cancer, and carcinoma in situ of uterine cervix
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis or on oral anti-vitamin K medication
* Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control from enrollment through 6 months following the end of treatment
* Patients who have received prior treatment with an mTOR inhibitor.
* Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, MD, Principal Investigator — University of Chicago
Locations (5):
- United States (5):
  - University of Chicago, Chicago, Illinois
  - Oncology/Hematology Associates, Peoria, Illinois
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - The University of North Carolina at Chapel Hill, Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina

REFERENCES:
- [Result] Chen JL, Appelbaum DE, Kocherginsky M, Cowey CL, Rathmell WK, McDermott DF, Stadler WM. FDG-PET as a predictive biomarker for therapy with everolimus in metastatic renal cell cancer. Cancer Med. 2013 Aug;2(4):545-52. doi: 10.1002/cam4.102. Epub 2013 Jul 10. PMID 24156027
- See also: Study results publication available through PMC — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3799289/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 patients started trial between December, 2007 and June, 2010 at 5 clinical sites. . A total of 63 patients signed consent, (1 withdrew consent, 2 failed screening)
Pre-assignment Details: This is a single-arm trial.
Groups:
- Everolimus: All patients were to receive 10mg everolimus (RAD001) daily.
Period: Evaluable for Primary Endpoint
Arm/Group | Everolimus
Started | 60 (60 patients started trial)
Completed | 50 (Evaluable for primary endpoint)
Not Completed | 10
Not completed — Did not complete 2d CT scan | 3
Not completed — Worsening performance status | 2
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 1
Period: Evaluable for Secondary Endpoint
Arm/Group | Everolimus
Started | 50
Completed | 48
Not Completed | 2
Not completed — Did not complete 2d FDG-PET scan | 2

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 35
Tumor Type [Number; unit: participants]
  Clear Cell | 36
  Papillary Cell | 4
  Chromophobe | 4
  Unclassified/Other | 6
Average SUVmax [Number; unit: participants] — The standardized uptake value (SUV) was calculated for each FDG-PET scan. The average of the maximum SUV (SUVmax) across all lesions (aveSUVmax) on the baseline scan was used to classify patients into low- and high-uptake. Low uptake group was defined as avgSUVmax <=4, and high uptake group was defined as avgSUVmax > 4.
  participants
    Low Uptake (avgSUVmax<=4) | 10
    High Uptake (avgSUVmax>4) | 40

OUTCOME MEASURES:

1. Primary Outcome: Relative Tumor Size Change Following 8 Weeks of Therapy.
Description: The primary objective is to determine whether high SUV uptake on FDG-PET is associated with greater tumor shrinkage. Tumor size is defined as the sum of unidimensional tumor measurements from standard CT imaging calculated according to RECIST criteria. Tumor size is measured at baseline and after eight weeks of therapy. Tumor shrinkage is the relative change (%) in tumor size from baseline.
Time Frame: 8 weeks
Population: 50 patients were evaluable for response and had a baseline FDG-PET scan.
Measure: Mean (Full Range); unit: Percent change from baseline
Groups:
- Low Uptake: Low uptake FDG-PET is defined as avgSUVmax<=4; avgSUVmax is the average across all measured lesions of each lesion's maximum SUV (SUV is the "standardized uptake value") .
- High Uptake: High uptake of FDG-PET defined as avgSUVmax>4; avgSUVmax is the average across all measured lesions of each lesion's maximum SUV (SUV is the "standardized uptake value") .
Arm/Group | Low Uptake | High Uptake
Number analyzed (Participants) | 10 | 40
Percent change from baseline | 1.4 [-31.7 to 17.3] | -0.57 [-32.7 to 35.9]
Statistical Analysis 1: Comparison: Low Uptake vs High Uptake; Relative changes in tumor size were log-transformed to satisfy the normality assumption; Test type: Superiority or Other; p = 0.69, t-test, 2 sided; Relative changes in tumor size were log-transformed to satisfy the normality assumption for the t-test; Mean Difference (Net) = 1.9, 95% CI 2-sided [-9.3 to 13.23] — Mean difference is the difference between Low and High SUV uptake groups in tumor size percent (%) change from baseline, and is reported on the raw scale. Tumor size changes were log-transformed for the t-test

2. Secondary Outcome: Percent Change in FDG-PETUptake Following 2 Weeks of Therapy
Description: The secondary objective was to explore whether an early change in FDG-PET uptake is associated with tumor shrinkage. Change in FDG-PET uptake was calculated using the baseline and 2-week FDG-PET scans.
Time Frame: 2 weeks
Population: Patients evaluable for tumor response at 8 weeks who also had both the baseline and 2-week FDG-PET scans.
Measure: Mean (Full Range); unit: % change in avgSUVmax at 2 weeks
Groups:
- Patients Evaluable for Secondary Outcome: Patients who had two FDG-PET scans completed, one at baseline and one after 2 weeks of treatment, were evaluable for secondary outcome.
Arm/Group | Patients Evaluable for Secondary Outcome
Number analyzed (Participants) | 48
% change in avgSUVmax at 2 weeks | -29.7 [-75.3 to 0]
Statistical Analysis 1: Comparison: Patients Evaluable for Secondary Outcome; The relationship between early changes in SUV uptake (from baseline to 2 weeks) and tumor size changes (from baseline to 8 weeks) were examined using linear regression models. Tumor size change was log-transformed to satisfy the normality assumption; Test type: Superiority or Other; p = 0.013, Regression, Linear; Tumor size change (outcome variable) was log-transformed to satisfy the normality assumption; Slope = 0.0028, 95% CI 2-sided [0.00063 to 0.004997], Standard Error of Mean .00109 — Outcome was log(tumor size at 8 weeks/tumor size at baseline), and the predictor was the early change in aveSUVmax [(aveSUVmax at 2 weeks - aveSUVmax at baseline)/aveSUVmax at baseline] x 100%

ADVERSE EVENTS:
Description: These results are based on n=56 patients who were evaluable for toxicity (all patients started treatment but 4 had missing data).
Groups:
- Everolimus: All patients were to receive 10mg everolimus (RAD001) daily.
  These results are based on n=56 patients who were evaluable for toxicity.
Arm/Group | Everolimus
Serious Adverse Events (participants affected / at risk) | 6/56
Other Adverse Events (participants affected / at risk) | 55/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=56)
Creatinine increased (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=56)
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 6
Diarrhea (Gastrointestinal disorders) | 21
Dizziness (Nervous system disorders) | 5
Dry mouth (Gastrointestinal disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19
Ear, nose and throat examination abnormal (Ear and labyrinth disorders) | 25
Edema limbs (General disorders) | 16
Fatigue (General disorders) | 40
Fever (General disorders) | 8
Flatulence (Gastrointestinal disorders) | 3
General symptom (General disorders) | 6
Headache (Nervous system disorders) | 10
Hemoglobin decreased (Investigations) | 23
Hemorrhage nasal (General disorders) | 5
Hypercholesterolemia (Investigations) | 21
Hyperglycemia (Metabolism and nutrition disorders) | 22
Hyperkalemia (Metabolism and nutrition disorders) | 9
Hypertriglyceridemia (Metabolism and nutrition disorders) | 24
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 11
Insomnia (Psychiatric disorders) | 6
Joint pain (Musculoskeletal and connective tissue disorders) | 3
Leukocytes (Investigations) | 5
Lymphopenia (Investigations) | 6
Mucositis oral (Gastrointestinal disorders) | 4
Nail changes (Skin and subcutaneous tissue disorders) | 5
Nausea (Gastrointestinal disorders) | 21
Neurological disorder NOS (Nervous system disorders) | 3
Pain (General disorders) | 8
Pain - Other (General disorders) | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Platelet count decreased (Investigations) | 10
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 5
Pulmonary - Other(specify) (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 15
Rash desquamating (Skin and subcutaneous tissue disorders) | 10
Rigors/chills (General disorders) | 4
Sinus tachycardia (Cardiac disorders) | 3
Taste alteration (General disorders) | 8
Urinary frequency (Renal and urinary disorders) | 4
Urinary tract infection (Infections and infestations) | 3
Vomiting (Gastrointestinal disorders) | 7
Weight loss (Investigations) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less